CLINICAL TRIAL: NCT00103454
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter, Study to Evaluate the Efficacy and Safety of Once-Daily, Intranasal Administration of GW685698X Aqueous Nasal Spray 100mcg for 4 Weeks in Adult and Adolescent Subjects (12 Years of Age and Older) With Perennial Allergic Rhinitis (PAR)
Brief Title: A Study To Evaluate The Efficacy And Safety Of A Once-Daily Investigational Nasal Spray In Adults And Adolescents With Perennial Allergic Rhinitis (PAR).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FFR30002
Record Dates: First submitted 2005-02-08; First posted 2005-02-09 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: allergic rhinitis; GW685698X; Perennial Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: GW685698X

INTERVENTIONS:
Drug: GW685698X

SUMMARY:
The primary objective of this study is to compare the efficacy and safety of GW685698X 100mcg once daily (QD) aqueous nasal spray with vehicle placebo nasal spray in adult and adolescent subjects (12 years of age and older) with perennial allergic rhinitis (PAR).

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy and Safety of Once-Daily, Intranasal Administration of GW685698X Aqueous Nasal Spray 100mcg for 4 Weeks in Adult and Adolescent Subjects (12 years of age and older) with Perennial Allergic Rhinitis (PAR)

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of perennial allergic rhinitis (PAR).
* Must comply with study procedures and be literate.

Exclusion criteria:

* Significant concomitant medical conditions.
* Use of corticosteroids.
* Use of allergy medications and some other medications during the study.
* Current tobacco use.
* Clinically significant abnormal ECG or laboratory abnormality.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2005-01; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline over the entire treatment period in daily, reflective total nasal symptom scores. Subjects complete diaries twice daily (every 12 hours) reporting the severity of their PAR symptoms.

SECONDARY OUTCOMES:
Mean change from baseline over the entire treatment period in AM, pre-dose, instantaneous total nasal symptom scores. The subject completes an overall evaluation of response to therapy during the last clinic visit.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (46):
- United States (40):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Vero Beach, Florida
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Lilburn, Georgia
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Portland, Maine
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, North Andover, Massachusetts
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Ocean City, New Jersey
  - GSK Investigational Site, Summit, New Jersey
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Lake Oswego, Oregon
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, New Braunfels, Texas
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, South Burlington, Vermont
  - GSK Investigational Site, West Allis, Wisconsin
- Canada (6):
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Nathan R, Berger W, Yang W, Cheema A, Silvey MJ, Wu W, Faris M, Philpot E. Once daily fluticasone furoate* nasal spray (FFNS), a novel enhanced affinity steroid, provides 24-hour relief for the nasal symptoms of perennial allergic rhinitis (PAR) J Allergy
- [Derived] Nathan RA, Berger W, Yang W, Cheema A, Silvey M, Wu W, Philpot E. Effect of once-daily fluticasone furoate nasal spray on nasal symptoms in adults and adolescents with perennial allergic rhinitis. Ann Allergy Asthma Immunol. 2008 May;100(5):497-505. doi: 10.1016/S1081-1206(10)60477-2. PMID 18517084
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: FFR30002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: FFR30002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: FFR30002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: FFR30002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: FFR30002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: FFR30002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: FFR30002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register